CLINICAL TRIAL: NCT03969875
Title: Comparison of the Analgesic Efficacy of a Single Shot Interscalene Block With Liposomal Bupivacaine to Bupivacaine With Dexamethasone as an adjuvant-a Randomized Controlled Trial
Brief Title: Comparison of Analgesic Efficacy Between of Interscalene Block With Liposomal Bupivacaine With Bupivacaine and Dexamethasone
Status: Completed | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Meg Rosenblatt, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 18-1264
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Results first posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-04

CONDITIONS: Total Shoulder Arthroplasty; Shoulder Osteoarthritis
Keywords: Liposomal bupivacaine; Dexamethasone; Interscalene catheter; Interscalene single shot
MeSH Terms: interventions — Dexamethasone; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | Unapproved Device: Yes

ARMS (3):
- Interscalene catheter (Active Comparator): Interscalene catheter 0.5 % bupivacaine 15cc with rescue catheters attached to a PCA pump with bupivacaine infusion at 6cc /hour.
  Interventions: Device: Interscalene catheter; Drug: Bupivacaine
- Interscalene single shot with liposomal bupivacaine (Experimental): Liposomal bupivacaine 10cc of exparel with 0.5% bupivacaine 5cc, total 15cc with rescue catheter attached to a PCA pump with normal saline at 6cc/hour infusion.
  Interventions: Drug: Liposomal bupivacaine
- Interscalene with bupivacaine and dexamethasone (Experimental): Interscalene single shot with bupivacaine and dexamethasone as adjuvant 0.5% bupivacaine 14cc with 1 cc of 4mg dexamethasone, total 15cc with rescue catheter attached to a PCA pump with normal saline at 6cc/hour infusion.
  Interventions: Drug: Dexamethasone; Drug: Bupivacaine

INTERVENTIONS:
Device: Interscalene catheter — rescue catheters attached to a PCA pump
  Arms: Interscalene catheter
Drug: Liposomal bupivacaine — 10 cc
  Other Names: Exparel
  Arms: Interscalene single shot with liposomal bupivacaine
Drug: Dexamethasone — 1 cc of 4mg
  Arms: Interscalene with bupivacaine and dexamethasone
Drug: Bupivacaine — 0.5% bupivacaine
  Arms: Interscalene catheter; Interscalene with bupivacaine and dexamethasone

SUMMARY:
Pain management after shoulder surgeries poses a unique challenge to the surgeon as well as the anesthesiologist. Regional anesthesia in the form of interscalene approach to the brachial plexus as an adjunct to general anesthesia or as a sole primary technique comes to one's rescue. Interscalene block either as single shot or as a catheter is an established modality for effective analgesia which facilitates early mobilization helping in physical therapy and early discharge.

With the help of local anesthetic injected as a single shot, analgesia usually lasts less than 24 hours. Recent research in regional anesthesia is advancing towards adjuvants which will prolong the duration of local anesthesia. This has introduced the concept of "multimodal perineural analgesia (MMPNA)" whereby multiple agents with differing mechanisms of action are used with the goal of providing perineural analgesia while avoiding exposure to high and potentially toxic levels of individual agents. Some of the commonly used adjuvants in clinical studies are fentanyl, buprenorphine, morphine, tramadol, magnesium, epinephrine, ketamine, non-steroidal anti-inflammatory drug (NSAID), midazolam, parecoxib, ketorolac, clonidine, dexmedetomidine, dexamethasone, neostigmine and potassium. They find a distinct place in wide spread clinical practice as an off-label use.

Steroids have a long history of safe use in epidural space for treatment of radicular pain due to nerve irritation. Dexamethasone is used routinely as a part of anti- emetic prophylaxis and anti-inflammatory effect. Methyl prednisone was the first steroid to be used as an adjuvant. Dexamethasone was first used as an adjuvant in 2003.

It has been hypothesized that steroids induce a degree of vasoconstriction, thereby reducing local anesthetic absorption, tend to have an opioid sparing effect. Another theory suggests that it increases the activity of inhibitory potassium channels on nociceptive C-fibers (via glucocorticoid receptors), thus decreasing their activity.

Several studies have demonstrated promising results with the use of 8mg of perineural dexamethasone. No neuronal injury has been reported in in vivo studies. Though there are several studies which report usage of dexamethasone in varying doses of 2mg to 8mg, the optimal effective dose of dexamethasone as an adjuvant for nerve block remains unknown. Some studies have suggested perineural is more effective than IV as an adjuvant .

Liposomal bupivacaine, a formulation where bupivacaine is encapsulated into multivesicular liposomes, making it a slow and controlled release from the liposomes, was originally indicated for wound infiltration at the surgical site to provide post-surgical analgesia. Studies have demonstrated efficacy up to 24 hours in femoral nerve block in total knee arthroplasty. Recent approval of liposomal bupivacaine in interscalene block for shoulder surgeries by FDA opens an arena unexplored in the world of regional anesthesia.

Current opioid epidemic, a crisis in health care forces healthcare providers to consider alternate analgesic modalities without compromising patient comfort. Regional anesthesia has revolutionized peri-operative pain management by avoiding opioids and their side effects. Use of adjuvants to the current regional techniques holds promise in postsurgical analgesia.

The researchers propose to compare the analgesic efficacy of liposomal bupivacaine to bupivacaine with dexamethasone as an adjuvant in interscalene block with catheters for shoulder surgeries. Till date, there is not a single study comparing the three in current literature.

DETAILED DESCRIPTION:
There have been several studies demonstrating efficacy of dexamethasone in prolonging the analgesic effect when administered both perineurally and intra-venously as an adjuvant to local anesthesia demonstrating a dose effect relationship. Liposomal bupivacaine has shown promising results in total knee arthroplasty and there are a limited number of studies demonstrating efficacy in total shoulder arthroplasty.

If by comparing dexamethasone as an adjuvant to bupivacaine and liposomal formulation is deciphered, it can help in avoiding costs associated with liposomal bupivacaine extending post-operative analgesia avoiding narcotics and reducing health care costs. And comparing the two to the standard catheters helps us understand if they have a role in pain management in the future.

ELIGIBILITY:
Inclusion Criteria:

* All patients between age 18-80 years undergoing elective primary total shoulder arthroplasty procedure.
* All patients who speak read and understand English will be included for follow up purposes.

Exclusion Criteria:

* Patient refusal
* ASA 5
* presence of coagulopathy
* severe lung disease
* contralateral diaphragmatic palsy
* insulin-dependent diabetes
* hepatic disease/failure
* kidney disease/failure
* pregnancy
* chronic opioid use (defined as opioid use for >3 months), or allergy to any of the study medications.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-08-18 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2022-04-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vandepitte C, Kuroda M, Witvrouw R, Anne L, Bellemans J, Corten K, Vanelderen P, Mesotten D, Leunen I, Heylen M, Van Boxstael S, Golebiewski M, Van de Velde M, Knezevic NN, Hadzic A. Addition of Liposome Bupivacaine to Bupivacaine HCl Versus Bupivacaine HCl Alone for Interscalene Brachial Plexus Block in Patients Having Major Shoulder Surgery. Reg Anesth Pain Med. 2017 May/Jun;42(3):334-341. doi: 10.1097/AAP.0000000000000560. PMID 28157791
- [Background] Abdallah FW, Brull R. Facilitatory effects of perineural dexmedetomidine on neuraxial and peripheral nerve block: a systematic review and meta-analysis. Br J Anaesth. 2013 Jun;110(6):915-25. doi: 10.1093/bja/aet066. Epub 2013 Apr 15. PMID 23587874
- [Background] Bishop JY, Sprague M, Gelber J, Krol M, Rosenblatt MA, Gladstone J, Flatow EL. Interscalene regional anesthesia for shoulder surgery. J Bone Joint Surg Am. 2005 May;87(5):974-9. doi: 10.2106/JBJS.D.02003. PMID 15866958

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from 2018 to 2022
Pre-assignment Details: There were 155 eligible participants and 90 were randomized.
Period: Overall Study
Arm/Group | Interscalene Catheter | Interscalene With Bupivacaine and Dexamethasone | Interscalene Single Shot With Liposomal Bupivacaine
Started | 31 | 29 | 30
Completed | 24 | 24 | 24
Not Completed | 7 | 5 | 6
Not completed — did not receive allocated intervention | 3 | 3 | 4
Not completed — Protocol Violation | 4 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Interscalene Catheter | Interscalene With Bupivacaine and Dexamethasone | Interscalene Single Shot With Liposomal Bupivacaine | Total
Number analyzed (Participants) | 24 | 24 | 24 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.08 (6.23) | 71.75 (6.58) | 68 (8.50) | 69.61 (7.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 17 | 13 | 44
  Male | 10 | 7 | 11 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 3 | 10
  Not Hispanic or Latino | 22 | 19 | 21 | 62
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 5 | 3 | 12
  White | 18 | 13 | 17 | 48
  More than one race | 2 | 5 | 3 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0
Type of Shoulder Replacement [Count of Participants; unit: Participants]
  Anatomic | 10 | 13 | 12 | 35
  Reverse | 14 | 11 | 12 | 37
Side of Surgery [Count of Participants; unit: Participants]
  Right | 12 | 13 | 15 | 40
  Left | 12 | 11 | 9 | 32
The American Society of Anesthesiologists (ASA) Physical Status Classification System [Count of Participants; unit: Participants] — ASA I - A normal healthy patient
  ASA II - A patient with mild systemic disease without significant functional limitation
  ASA III - A patient with severe systemic disease with significant functional limitation
  Participants
    ASA I | 1 | 0 | 0 | 1
    ASA II | 8 | 18 | 12 | 38
    ASA III | 15 | 6 | 12 | 33
Current Smoker [Count of Participants; unit: Participants] | 0 | 2 | 2 | 4
Level of Education [Count of Participants; unit: Participants]
  Under High School | 1 | 1 | 1 | 3
  High School | 10 | 9 | 5 | 24
  Bachelor | 7 | 8 | 10 | 25
  Graduate | 6 | 6 | 8 | 20
Number of Participant Employed [Count of Participants; unit: Participants] | 13 | 3 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: Numerical Rating Score for Pain
Description: Numerical rating score for pain is assessed from 0 to 10, with 0 being no pain and 10 being worst pain.
Time Frame: at 6 hours, 12 hours, 18 hours, 24 hours, 36 hours, 48 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Interscalene With Bupivacaine and Dexamethasone: Interscalene single shot with bupivacaine and dexamethasone as adjuvant 0.5% bupivacaine 14cc with 1 cc of 4mg dexamethasone, total 15cc with rescue catheter attached to a PCA pump with normal saline at 6cc/hour infusion.
  Dexamethasone: 1 cc of 4mg Bupivacaine: 0.5% bupivacaine
Arm/Group | Interscalene Catheter | Interscalene With Bupivacaine and Dexamethasone | Interscalene Single Shot With Liposomal Bupivacaine
Number analyzed (Participants) | 24 | 24 | 24
score on a scale
  6 hours | 0.00 [0.00 to 2.25] | 0.00 [0.00 to 3.00] | 0.00 [0.00 to 1.00]
  12 hours | 0.00 [0.00 to 5.00] | 0.00 [0.00 to 2.25] | 2.00 [0.00 to 7.00]
  18 hours | 2.00 [000 to 4.25] | 5.50 [0.00 to 7.00] | 0.50 [0.00 to 2.50]
  24 hours | 2.50 [0.00 to 5.00] | 3.00 [0.00 to 6.25] | 2.00 [0.00 to 3.00]
  36 hours | 3.00 [0.00 to 5.00] | 2.00 [0.75 to 5.25] | 2.00 [1.00 to 5.00]
  48 hours | 2.00 [0.00 to 3.25] | 2.00 [0.75 to 5.00] | 2.50 [0.75 to 5.00]

2. Secondary Outcome: Time to First Analgesic Request
Description: Time to first analgesic request on Day 1
Time Frame: Day 1
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Interscalene Catheter | Interscalene With Bupivacaine and Dexamethasone | Interscalene Single Shot With Liposomal Bupivacaine
Number analyzed (Participants) | 24 | 24 | 24
hours | 1.50 [0.16 to 18.00] | 3.50 [0.00 to 12.00] | 2.19 [0.15 to 9.00]

3. Secondary Outcome: Total Narcotic Consumption
Description: Total narcotic consumption in mg morphine equivalents (MME) during hospital stay
Time Frame: hospital stay, up to 48 hours
Measure: Median (Inter-Quartile Range); unit: MME
Groups:
- Interscalene With Bupivacaine and Dexamethasone Bupivacaine: Interscalene single shot with bupivacaine and dexamethasone as adjuvant 0.5% bupivacaine 14cc with 1 cc of 4mg dexamethasone, total 15cc with rescue catheter attached to a PCA pump with normal saline at 6cc/hour infusion.
  Dexamethasone: 1 cc of 4mg Bupivacaine: 0.5% bupivacaine
Arm/Group | Interscalene Catheter | Interscalene With Bupivacaine and Dexamethasone Bupivacaine | Interscalene Single Shot With Liposomal Bupivacaine
Number analyzed (Participants) | 24 | 24 | 24
MME | 30.00 [12.50 to 65.25] | 21.05 [5.62 to 57.45] | 13.25 [0.00 to 33.95]

4. Secondary Outcome: Arm Weakness
Description: Arm weakness as assessed by flexion and extension at wrist -- total scale from 1 to 10, with 10 being most weakness
Time Frame: at 6 hours, 12 hours, 18 hours, 24 hours, 36 hours
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Interscalene Catheter | Interscalene With Bupivacaine and Dexamethasone | Interscalene Single Shot With Liposomal Bupivacaine
Number analyzed (Participants) | 24 | 24 | 24
score on a scale
  6 hours | 2.00 [1.00 to 2.00] | 2.00 [0.75 to 3.00] | 2.00 [0.75 to 2.00]
  12 hours | 2.00 [1.75 to 3.25] | 3.00 [2.00 to 4.00] | 4.00 [2.00 to 4.00]
  18 hours | 3.00 [2.00 to 4.00] | 4.00 [3.00 to 5.00] | 4.00 [3.00 to 5.00]
  24 hours | 4.00 [3.00 to 5.00] | 5.00 [4.75 to 5.00] | 5.00 [4.00 to 5.00]
  36 hours | 5.00 [4.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [4.75 to 5.00]

5. Secondary Outcome: Arm Numbness
Description: Arm numbness assessed by the sensation at deltoid area. Sensation total scale from 1 to 10, with higher number indicating most sensation.
Time Frame: at 6 hours, 12 hours, 18 hours, 24 hours, 36 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Interscalene Catheter | Interscalene With Bupivacaine and Dexamethasone | Interscalene Single Shot With Liposomal Bupivacaine
Number analyzed (Participants) | 24 | 24 | 24
score on a scale
  6 hours | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 2.00]
  12 hours | 2.00 [1.00 to 2.00] | 2.00 [0.75 to 3.00] | 2.00 [0.75 to 2.00]
  18 hours | 2.00 [1.00 to 2.00] | 2.00 [2.00 to 2.00] | 2.00 [2.00 to 2.00]
  24 hours | 2.00 [2.00 to 2.00] | 2.00 [2.00 to 2.00] | 2.00 [2.00 to 2.00]
  36 hours | 2.00 [2.00 to 4.00] | 3.00 [2.00 to 4.00] | 2.00 [2.00 to 4.00]

6. Secondary Outcome: Time of Analgesia Duration
Description: The duration for which the patient has no pain on Day 1
Time Frame: Day 1
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Interscalene Catheter | Interscalene With Bupivacaine and Dexamethasone | Interscalene Single Shot With Liposomal Bupivacaine
Number analyzed (Participants) | 24 | 24 | 24
hours | 6.00 [1.50 to 17.00] | 11.00 [5.75 to 15.75] | 8.00 [5.00 to 16.50]

7. Secondary Outcome: Time of Motor Recovery
Description: Time of motor recovery on Day 1
Time Frame: Day 1
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Interscalene Catheter | Interscalene With Bupivacaine and Dexamethasone | Interscalene Single Shot With Liposomal Bupivacaine
Number analyzed (Participants) | 24 | 24 | 24
hours | 12.00 [10.00 to 24.00] | 14.00 [10.00 to 18.00] | 12.00 [6.75 to 18.00]

8. Secondary Outcome: Sensory Intact
Description: Sensory testing by using pinprick in the region of C5 dermatome. Scale from 1 to 10, with higher score indicating more sensation.
Time Frame: at 6 hours, 12 hours, 18 hours, 24 hours, 36 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Interscalene Catheter | Interscalene With Bupivacaine and Dexamethasone | Interscalene Single Shot With Liposomal Bupivacaine
Number analyzed (Participants) | 24 | 24 | 24
score on a scale
  6 hours | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  12 hours | 2.00 [1.00 to 2.00] | 2.00 [1.00 to 2.00] | 2.00 [1.00 to 2.00]
  18 hours | 2.00 [1.00 to 2.00] | 2.00 [1.00 to 2.00] | 2.00 [1.00 to 2.00]
  24 hours | 2.00 [2.00 to 2.00] | 2.00 [2.00 to 2.00] | 2.00 [2.00 to 2.00]
  36 hours | 2.00 [2.00 to 4.00] | 2.00 [2.00 to 4.00] | 2.00 [2.00 to 4.00]

9. Secondary Outcome: Hand Strength
Description: Hand strength assessed by using dynamometer, a device for measuring the amount of static force that can squeeze around a dynamometer, in kilograms.
Time Frame: at 6 hours, 12 hours, 18 hours, 24 hours, 36 hours
Measure: Median (Inter-Quartile Range); unit: kg
Arm/Group | Interscalene Catheter | Interscalene With Bupivacaine and Dexamethasone | Interscalene Single Shot With Liposomal Bupivacaine
Number analyzed (Participants) | 24 | 24 | 24
kg
  6 hours - Left hand | 16.90 [10.68 to 26.75] | 18.00 [12.00 to 20.80] | 16.35 [14.45 to 30.00]
  12 hours - Left hand | 13.50 [9.35 to 26.75] | 19.00 [12.00 to 21.00] | 16.85 [6.05 to 29.25]
  18 hours Left hand | 13.95 [9.17 to 26.55] | 16.50 [14.90 to 22.35] | 19.50 [8.45 to 31.25]
  24 hours - Left hand | 15.10 [10.00 to 26.75] | 19.00 [13.30 to 22.25] | 20.00 [9.75 to 35.25]
  36 hours - Left hand | 16.50 [9.80 to 26.50] | 20.00 [14.50 to 24.25] | 20.00 [11.50 to 35.25]
  6 hours - Right hand | 14.90 [8.75 to 23.95] | 13.50 [5.43 to 24.25] | 10.00 [2.00 to 22.70]
  12 hours - Right hand | 14.75 [9.00 to 22.00] | 14.50 [9.53 to 24.12] | 12.00 [4.57 to 22.65]
  18 hours - Right hand | 16.80 [9.90 to 22.75] | 16.35 [10.75 to 25.77] | 12.40 [7.35 to 21.83]
  24 hours - Right hand | 16.90 [10.68 to 26.75] | 19.30 [10.88 to 26.00] | 17.50 [8.75 to 25.25]
  36 hours - Right hand | 13.50 [9.35 to 26.75] | 20.50 [10.75 to 30.00] | 18.50 [10.00 to 25.75]

10. Secondary Outcome: PACU Length of Stay
Description: Post-anesthesia Care Unit length of stay in hours on Day 1
Time Frame: Day 1
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Interscalene Catheter | Interscalene With Bupivacaine and Dexamethasone | Interscalene Single Shot With Liposomal Bupivacaine
Number analyzed (Participants) | 24 | 24 | 24
hours | 2.7 [2.11 to 3.0] | 2.44 [2.0 to 3.0] | 3 [2.0 to 3.26]

11. Secondary Outcome: Hospital Length of Stay
Description: Length of stay for duration of hospital admission
Time Frame: up to 3 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Interscalene Catheter | Interscalene With Bupivacaine and Dexamethasone | Interscalene Single Shot With Liposomal Bupivacaine
Number analyzed (Participants) | 24 | 24 | 24
days | 2.75 [1.0 to 3.0] | 2 [1.0 to 2.5] | 1.75 [1.0 to 3.0]

12. Secondary Outcome: Number of Complication Events
Description: Number of complications - any associated complications like nausea, vomiting, dizziness, horner's syndrome, hoarseness and dyspnea
Time Frame: up to 3 days
Measure: Number; unit: events
Arm/Group | Interscalene Catheter | Interscalene With Bupivacaine and Dexamethasone | Interscalene Single Shot With Liposomal Bupivacaine
Number analyzed (Participants) | 24 | 24 | 24
events
  Nausea | 3 | 2 | 1
  Vomiting | 0 | 0 | 0
  Dizziness | 2 | 2 | 2
  Horners | 2 | 0 | 0
  Hoarseness | 1 | 3 | 0
  Dyspnea | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Quality of Sleep Rating
Description: Patient to rate their quality of sleep as good, average, or bad
Time Frame: average of 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Interscalene Catheter | Interscalene With Bupivacaine and Dexamethasone | Interscalene Single Shot With Liposomal Bupivacaine
Number analyzed (Participants) | 24 | 24 | 24
Participants
  Good | 12 | 9 | 7
  Average | 5 | 6 | 7
  Bad | 7 | 9 | 10

14. Secondary Outcome: Number of Participants With Patient's Satisfaction
Description: Number of Participants with Patient satisfaction. Patients were asked if they were satisfied.
Time Frame: during the hospital stay, up to 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Interscalene Catheter | Interscalene With Bupivacaine and Dexamethasone | Interscalene Single Shot With Liposomal Bupivacaine
Number analyzed (Participants) | 24 | 24 | 24
Participants | 16 | 16 | 16

15. Secondary Outcome: Change in Patient Reported Outcomes Measurement Information System (PROMIS)
Description: PROMIS global assessment assesses physical and mental activities of daily living scored from 0 (poor) to 5 (excellent) at first post-operative visit as compared to baseline. Each scale from 0-100, higher score indicates better health outcomes.
Time Frame: baseline and one week post-op
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Interscalene Catheter | Interscalene With Bupivacaine and Dexamethasone | Interscalene Single Shot With Liposomal Bupivacaine
Number analyzed (Participants) | 24 | 24 | 24
score on a scale
  Pre-Physical, baseline | 41.98 (9.88) | 42.42 (8.83) | 42.19 (9.26)
  Post-Physical, one week post-op | 44.44 (9.57) | 43.55 (9.52) | 45.15 (8.89)
  Pre-Mental, baseline | 50.00 (12.18) | 51.64 (11.01) | 51.44 (8.35)
  Post-Mental, one week post-op | 49.75 (11.51) | 52.14 (10.41) | 52.99 (6.93)

ADVERSE EVENTS:
Time Frame: average 48 hours
Arm/Group | Interscalene Catheter | Interscalene With Bupivacaine and Dexamethasone | Interscalene Single Shot With Liposomal Bupivacaine
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-25): https://cdn.clinicaltrials.gov/large-docs/75/NCT03969875/Prot_SAP_000.pdf